CLINICAL TRIAL: NCT02169583
Title: A Two Part, Phase I, Randomized, Placebo Controlled, Double Blind Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Repeat Escalating Doses of GSK1325756 Solution for Infusion, and Absolute Bioavailability Relative of an Oral Dose, in Healthy Adult Subjects Protocol 201022
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Repeat Escalating Doses of GSK1325756 Solution for Infusion, and Absolute Bioavailability Relative of an Oral Dose, in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201022
Record Dates: First submitted 2014-06-05; First posted 2014-06-23 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Infections, Respiratory Tract
Keywords: GSK1325756; Safety; Bioavailability; Pharmacokinetics
MeSH Terms: conditions — Respiratory Tract Infections | interventions — danirixin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Cohort 1) (Experimental): Approximately 8 subjects (6 Active, 2 Placebo) will be randomized to receive single escalating IV doses i.e.10 milligrams (mg), 25 mg and 100 mg, plus one oral 100 mg dose (on the last occasion) of GSK1325756 or matching placebo, with a 7-days washout between doses. Dose escalations will be based on review of PK and safety data from preceding dose level. The projected doses for each group are subject to modification based upon PK and safety data from preceding cohorts. Pharmacokinetic parameters will be reviewed from at least 4 active subjects from preceding dose before dose escalating to the next dose level. The maximum dose administered will be 100 mg. Additional subjects/Cohorts may be enrolled.
  Interventions: Drug: GSK1325756 Solution; Drug: GSK1325756 Solution Matching Placebo; Drug: GSK1325756 Tablet; Drug: GSK1325756 Tablet Matching Placebo
- Part B (Cohorts 2 and 3) (Experimental): Approximately 8 subjects (6 Active, 2 Placebo) per cohort will be randomized to receive escalating repeated IV doses of GSK1325756 or matching placebo (Cohort 2: 25 mg, Cohort 3: 50 mg) for 5 days. Repeated (BID) doses of GSK1325756 will begin the morning of Day 1 and continue through the morning of Day 5 (9 total doses). Dose escalations will be based on review of PK and safety data from preceding dose level. The projected doses for each group are subject to modification based upon PK and safety data from preceding cohorts. Pharmacokinetic parameters will be reviewed from at least 4 active subjects from preceding dose before dose escalating to the next dose level. The maximum dose administered will be 50 mg BID. Additional subjects/Cohorts may be enrolled.
  Interventions: Drug: GSK1325756 Solution; Drug: GSK1325756 Solution Matching Placebo

INTERVENTIONS:
Drug: GSK1325756 Solution — Solution containing 2 mg/mL GSK1325756 in sterile water for injection, to be administered intravenously.
Drug: GSK1325756 Solution Matching Placebo — Solution containing sterile water for injection matching GSK1325756 solution, to be administered intravenously.
Drug: GSK1325756 Tablet — A white film coated tablet containing 50 mg GSK1325756 to be administered orally.
  Arms: Part A (Cohort 1)
Drug: GSK1325756 Tablet Matching Placebo — A white film coated tablet matching GSK1325756 tablet, to be administered orally.
  Arms: Part A (Cohort 1)

SUMMARY:
This will be the first time GSK1325756 Solution for Infusion formulation that has been administered to humans. Prior studies have been performed with oral GSK1325756. The primary objectives of this study are to obtain information on the safety, tolerability, and pharmacokinetics (PK) of single and twice daily intravenous (IV) administration of GSK1325756 in healthy subjects. In Part A, single, escalating doses will be given in the same cohort of subjects after a seven day washout. In addition, the study will evaluate the absolute bioavailability of a single dose of the current oral tablet formulation as compared to the IV formulation in Part A. In Part B, twice daily (BID) intravenous dose administration will be given for 5 days (9 total doses) in two separate cohorts of subjects. Data from this study will provide understanding of the safety, tolerability, and PK of intravenously administered GSK1325756 twice daily to guide dose selection in future clinical studies in patients with viral respiratory tract infections

ELIGIBILITY:
Inclusion Criteria:

* Males/females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including (medical history, physical examination, laboratory tests and ECG). A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Body weight >=60 kilograms (kg) for men and >=45 kg for women; and Body Mass Index (BMI) within the range 19 to 32 kg/square meter (m^2) (inclusive).
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international unit (MIU)/milliliter (mL) and estradiol <40 picograms (pg)/mL (<147 picomoles [pmol]/liter [L]) is confirmatory].
* Male subjects with female partners of child-bearing potential must agree to use one of the acceptable contraception methods. This criterion must be followed from the time of the first dose of study medication until 90 days following the last dose.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on a single ECG obtained over a brief recording period: corrected QT interval (QTc) <450 milliseconds (msec); or QTc <480 msec in subjects with Bundle Branch Block.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* Part A only: Subjects currently or likely to take antacids (H2 receptor antagonists, proton pump inhibitors [PPI] blockers, etc.) at any point during the study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Urinary cotinine levels indicative of smoking history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Pregnant females as determined by positive (serum or urine) human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Subjects with a peripheral blood neutrophil count at the screening visit <2 x 10^9/L.
* Subjects with a history of renal disease or subjects with an abnormal urinalysis (confirmed on repeat) suggesting the possibility of renal disease (e.g. proteinuria).
* Subjects with a serum creatinine at the screening visit >1 x ULN.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2014-08-28 (Actual); Study Completion 2014-08-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) | Part A and Part B: from Day -1 until 7 to 10 days post-last dose
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Changes over time in clinical laboratory evaluations from pre-dose values | Part A and Part B: from Day -1 until 7 to 10 days post-last dose
  Clinical laboratory assessments will include hematology, clinical chemistry, urinalysis parameters
Changes over time in vital signs from pre-dose values | Part A and Part B: from Day -1 until 7 to 10 days post-last dose
  Vital sign measurements will include systolic and diastolic blood pressure and pulse rate
Changes over time in electrocardiogram (ECG) parameters from pre-dose values | Part A and Part B: from Day -1 until 7 to 10 days post-last dose
  12-lead ECGs will be obtained at each timepoint
GSK1325756 PK parameters following single dose administration in Part A and on Day 1 of Part B | Part A: Pre-dose, 0.5 hour (hr), 1hr (end of infusion/post oral dose), 1.5, 2, 3, 4, 8, 12, 24hrs post-dose in each treatment period.
  PK parameters will include area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time [AUC(0-infinity)], area under the concentration-time curve from time zero (pre-dose) to time t [AUC(0-t)], area under the concentration-time curve from time zero (pre-dose) to 24 hours [AUC(0-24)], maximum observed concentration (Cmax), time to maximum observed concentration (tmax), observed concentration at 24 hours post-dose (C24), terminal half-life (t1/2), time of last measurable concentration (tlast), clearance (CL) and volume of distribution (Vz)
GSK1325756 PK parameters following repeat dose administration (Part B, Day 5) | Part B: Day 5 at pre-dose, 0.5, 1hr (end of infusion), 1.5, 2, 3, 4, 8, 12 and 24 hrs post-dose
  PK parameters will include area under the concentration-time curve from time zero (pre-dose) to the end of the dosing interval [AUC(0-tau)], concentration at the end of the dosing interval (Ctau), Cmax, tmax, t1/2, Volume of distribution at steady-state (Vdss), and oral clearance (CL/F)

SECONDARY OUTCOMES:
GSK1325756 PK parameters following single and repeat IV dose administration to assess dose proportionality | Part A: Pre-dose, 0.5hr, 1hr (end of infusion/post oral dose), 1.5, 2, 3, 4, 8, 12, 24hrs post-dose. Part B: Day 1 and Day 5: pre-dose, 0.5, 1hr (end of infusion), 1.5, 2, 3, 4, 8, 12 and (Day 5 only) 24 hrs post-dose. Day 2-4: pre-dose (each dose)
  PK parameters will include AUC(0-infinity), AUC(0-t), Cmax, and C24 following single IV dose administration (Part A) and AUC(0-tau), Ctau, and Cmax following repeated IV dose administration (Part B)
GSK1325756 PK parameters following single IV and oral dose administration of a given dose of GSK1325756 (Part A) to determine the absolute bioavailability | Part A: Pre-dose, 0.5hr, 1hr (end of infusion/post oral dose), 1.5, 2, 3, 4, 8, 12, 24hrs post-dose
  PK parameters will include AUC(0-infinity), AUC(0-t), Cmax and tmax
GSK1325756 accumulation ratio | Part A: Pre-dose, 0.5hr, 1hr (end of infusion/post oral dose), 1.5, 2, 3, 4, 8, 12, 24hrs post-dose Part B: Day 1 and Day 5: pre-dose, 0.5, 1hr (end of infusion), 1.5, 2, 3, 4, 8, 12 and (Day 5 only) 24 hrs post-dose. Day 2-4: pre-dose (each dose)
  GSK1325756 AUC(0-tau), Cmax, and Ctau on the last day of dosing will be compared to area under the concentration-time curve from time zero (pre-dose) to 12 hours [AUC(0-12)], Cmax, and observed concentration at 12 hours post-dose (C12) on Day 1 to estimate accumulation ratio
GSK1325756 time invariance | Part A: Pre-dose, 0.5hr, 1hr (end of infusion/post oral dose), 1.5, 2, 3, 4, 8, 12, 24hrs post-dose Part B: Day 1 and Day 5: pre-dose, 0.5, 1hr (end of infusion), 1.5, 2, 3, 4, 8, 12 and (Day 5 only) 24 hrs post-dose. Day 2-4: pre-dose (each dose)
  GSK1325756 AUC(0-tau) on the last day of dosing in Part B, will be compared to AUC(0-infinity) on Day 1 of Part A to evaluate time invariance
GSK1325756 Pre-dose concentrations (C12/Ctau) on Day 2 through 4 | Part B: Day 2 to Day 4 (pre-dose; each dose)
  GSK1325756 Pre-dose concentrations on Day 2 through 4 will be used to assess the achievement of steady state of GSK1325756 following repeat administration (Part B)
Correlation between PK parameters and various safety parameters, if appropriate | Part A and Part B: from Day -1 until 7 to 10 days post-last dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 201022 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201022?search=study&search_terms=201022#rs
- Available data/document: Dataset Specification: 201022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register